CLINICAL TRIAL: NCT00462501
Title: A Pilot Study of Neoadjuvant Chemotherapy With Selective Use of Radiation for Locally Advanced Rectal Cancer
Brief Title: Combination Chemotherapy and Bevacizumab With or Without Radiation Therapy in Treating Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-021; P30CA008748 (NIH); MSKCC-07021
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin; Radiotherapy

ARMS (1):
- Chemotherapy and Bevacizumab With or Without Radiation (Experimental): FOLFOX/Bevacizumab will be given for 4 cycles over 8 weeks; FOLFOLX6 without Bevacizumab will be given for an additional 2 cycles over 4 weeks. Oxaliplatin will be given on Day 1 of each cycle over 2 hours at 85 mg/m2 IV. Leucovorin will be given Day 1 of each cycle over 2 hours at 400 mg/m2 IV. Fluorouracil will be given on Day 1 of each cycle at 400 mg/m2 IVP, then Fluorouracil will be given at 1200 mg/m2 IVCI over Day 1 and 2. Bevacizumab will be given at 5mg/kg over 10 minutes on day 1. Patients will undergo re-staging within 3 weeks of completing their 6th cycle of FOLFOX. If the reassessment reveals that there has been no disease progression as compared to the pre-treatment evaluation and the patient remains a candidate for an R0 resection. If the surgical oncologist's reassessment is that the patient is not a candidate for an R0 resection, the patient will proceed to standard pre-operative radiation with synchronous infusional 5-fluorouracil.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of rectal cancer by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy and bevacizumab together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy and bevacizumab with or without radiation therapy works in treating patients with locally advanced rectal cancer

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether neoadjuvant chemotherapy comprising oxaliplatin, fluorouracil, leucovorin calcium (FOLFOX), and bevacizumab can be substituted for pelvic radiotherapy without compromising R0 resection rates in patients with locally advanced rectal cancer.

Secondary

* Determine whether a 3-year local recurrence rate of ≤ 10% can be achieved in patients treated with this regimen.
* Determine the proportion of patients who achieve a complete pathologic response after treatment with this regimen.

OUTLINE: This is a non-randomized, open-label, pilot study.

* Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV over 10 minutes on day 1 and fluorouracil IV continuously over 48 hours on days 1 and 2 in weeks 1, 3, 5, and 7. Patients then receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 48 hours on days 1 and 2 in weeks 9 and 11. Treatment continues in the absence of disease progression or unacceptable toxicity.

Within 3 weeks after completion of neoadjuvant chemotherapy, patients undergo restaging evaluation. Patients with no evidence of disease progression by endorectal ultrasound (ERUS), pelvic MRI, and CT scan of the chest/abdomen AND who remain candidates for R0 resection may proceed directly to surgical resection within 4-6 weeks after completion of neoadjuvant chemotherapy. Patients with progressive disease who are not candidates for an R0 resection, proceed to neoadjuvant chemoradiotherapy.

* Neoadjuvant chemoradiotherapy: Patients undergo pelvic radiotherapy 5 days a week and receive concurrent fluorouracil IV continuously for 5½ weeks. Within 4-7 weeks after completion of chemoradiotherapy, patients undergo surgical resection.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or pathologically confirmed adenocarcinoma of the rectum

  * Clinical stage T1, N1; T2, N1; T3, N0; or T3, N1 by endorectal ultrasonography (ERUS)

    * No bulky N2 disease by either ERUS or MRI
    * No primary fixed or unresectable (clinical stage T4) rectal cancer or recurrent colorectal cancer limited to the pelvis

      * Primary unresectable rectal cancer is defined as a primary rectal tumor which on the basis of either physical exam, ERUS or pelvic MRI is deemed to be adherent or fixed to adjacent pelvic structures
* Must be a candidate for all of the following:

  * Neoadjuvant chemoradiotherapy
  * Systemic therapy with fluorouracil, leucovorin calcium, oxaliplatin (FOLFOX), and bevacizumab
  * Complete surgical resection via low anterior resection prior to administration of any therapy
* No low-lying tumors deemed to require an abdominal perineal resection
* No large or bulky tumors that require a diverting colostomy or placement of an endorectal stent prior to treatment initiation
* No clinical evidence of metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count > 150,000/mm^3
* Hemoglobin > 8.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study therapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No arterial thrombotic event within the past 6 months, including stable or unstable angina, myocardial infarction (MI), or cerebral vascular accident (CVA)

  * Deep venous thrombosis, pulmonary embolus, MI, CVA, atrial fibrillation, or any other conditions occurring more than 6 months ago allowed provided patient is on stable doses of anticoagulant therapy
* No other medical or psychiatric condition or disease that would preclude study therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or surgery for rectal cancer
* No prior pelvic radiotherapy
* No other concurrent experimental therapy, including any of the following:

  * Chemotherapy
  * Radiotherapy
  * Hormonal therapy
  * Antibody therapy
  * Immunotherapy
  * Gene therapy
  * Vaccine therapy
  * Angiogenesis inhibitors
  * Matrix metalloprotease inhibitors
  * Thalidomide
  * Anti-vascular endothelial growth factor/Flk-1 monoclonal antibody
  * Any other experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Karyn A. Goodman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Martin Weiser, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy and Bevacizumab With or Without Radiation
Started | 35
Completed | 30
Not Completed | 5
Not completed — Not treated | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy and Bevacizumab With or Without Radiation
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response
Description: This will be assessed on the basis of the surgical pathology report.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Chemotherapy and Bevacizumab With or Without Radiation
Number analyzed (Participants) | 30
participants
  Complete Response | 8
  Partial Response | 21
  Unknown | 1

ADVERSE EVENTS:
Arm/Group | Chemotherapy and Bevacizumab With or Without Radiation
Serious Adverse Events (participants affected / at risk) | 11/35
Other Adverse Events (participants affected / at risk) | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and Bevacizumab With or Without Radiation (N=35)
Cardiac Arrhythmia, other (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infection, other (Infections and infestations) | 1 (1)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and Bevacizumab With or Without Radiation (N=35)
Alanine aminotransferase increased (Investigations) | 3 (6)
Aspartate aminotransferase increase (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9)
Alkaline phosphatase increase (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (12)
Constipation (Gastrointestinal disorders) | 2 (3)
Creatinine increase (Investigations) | 3 (4)
Fatigue (General disorders) | 4 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (53)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 17 (94)
White blood cell decreased (Investigations) | 14 (23)
Lipase increased (Investigations) | 2 (7)
Lymphocyte count decreased (Investigations) | 10 (17)
Mucositis-Oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (8)
Neutrophil count decreased (Investigations) | 19 (42)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes